CLINICAL TRIAL: NCT05999851
Title: Multiparametric Assessment of Maternal Vascular Function as a New Diagnostic and Prognostic Tool for Hypertensive Disorders of Pregnancy and Preeclampsia - EDIPE Study
Brief Title: Multiparametric Assessment of Maternal Vascular Function in the Prediction of Hypertensive Disorders of Pregnancy
Acronym: EDIPE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Collaborators: University of Bologna (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 346/2023/Oss/AOUBo
Record Dates: First submitted 2023-06-15; First posted 2023-08-21 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-11

CONDITIONS: Preeclampsia; Hypertensive Disorder of Pregnancy
Keywords: Preeclampsia; Hypertensive Disorders of Pregnancy; Hypertension; Obstetric Medicine; Cardio-Obstetrics; Cardiovascular outcomes; Pregnancy complications; Arterial Stiffness; Endothelial Glycocalyx; Endothelial dysfunction; Uric Acid; Oxidative stress; Xanthine oxidase; Lipids
MeSH Terms: conditions — Pre-Eclampsia; Toxemia; Hypertension; Pregnancy Complications

STUDY DESIGN:
Intervention Model Description: The study is a single group study (Principal Arm) with a sub-group of participants undergoing additional experimental analyses. The additional analyses will be performed in participants who will develop hypertensive disorders of pregnancy and matched (age and body mass index before conception) controls with healthy pregnancies.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Principal arm (Experimental): The entire cohort of participants will undergo all experimental procedures. Participants who will develop hypertensive disorders of pregnancy and matched participants with healthy pregnancies will also undergo serum endothelial and angiogenic markers assessment.
  Interventions: Device: Arterial applanation tonometry; Device: In vivo endothelial glycocalyx measurement; Diagnostic Test: Serum markers of angiogenesis and endothelial dysfunction; Diagnostic Test: Blood chemistry test; Diagnostic Test: Serum xanthine oxidase activity

INTERVENTIONS:
Device: Arterial applanation tonometry — Arterial applanation tonometry will be performed at the carotid and femoral level by the PulsePen device (Software WPulsePen version 2.3.1, DiaTecne, Milan, Italy), while the subject is lying in the horizontal position and after 5 minutes of rest.
  Other Names: PulsePen; Arterial stiffness measurement; Pulse wave velocity assessment
Device: In vivo endothelial glycocalyx measurement — The in vivo microscopy (GlycoCheck system) is performed in the sublingual capillaries during the morning, with the participant sitting on a chair. The sublingual capillaries are visualized using an SDF video microscope (Capiscope handheld, KK Research technology Ltd).
  Other Names: Glycocheck; Sidestream dark field microscopy
Diagnostic Test: Serum markers of angiogenesis and endothelial dysfunction — ELISA assays to measure serum circulating markers of angiogenesis and endothelial dysfunction (ANG-1, ANG-2, ET-1, ICAM-1 and VCAM-1).
  Other Names: ANG-1; ET-1; ICAM-1; VCAM-1; ANG-2
Diagnostic Test: Blood chemistry test — Immunochemistry analysis of serum levels of uric acid, total cholesterol, LDL-cholesterol, HDL-cholesterol, Triglycerides, Lipoprotein (a)
Diagnostic Test: Serum xanthine oxidase activity — Serum xanthine oxidase (XO) activity will be assessed in blood samples measuring the ability of XO to produce uric acid

SUMMARY:
The present study is a single-centre prospective study that will enrol pregnant women during their first trimester of pregnancy (11+0 - 13+6 weeks of gestation).

During pregnancy, women will undergo standard clinical evaluation and management. During the two study visits (enrollment and 24+0 - 27+6 weeks of gestation) the investigators will perform arterial tonometry (Pulsepen) and in vivo darkfield microscopy (Glycocheck) to evaluate endothelial and vascular function. A urine sample and a blood sample for specific study analyses on metabolic profile, endothelial and angiogenic markers will be collected. Pregnancy outcomes will be collected at delivery and five years after delivery all the participants will be interview to collect long-term cardiovascular outcomes. Serum endothelial and angiogenic markers will be evaluated only in participants who will develop hypertensive disorders of pregnancy and in an equal number of controls matched for age and body mass index at the time of conception.

DETAILED DESCRIPTION:
Primary aim:

To determine the role of the combination of arterial tonometry and endothelial glycocalyx measurement in predicting the risk of developing hypertensive disorders in pregnancy.

Secondary aims:

* To determine the association between circulating markers of angiogenesis and endothelial dysfunction (ANG-1, ANG-2, ET-1, ICAM-1 and VCAM-1) and the development of hypertensive disorders of pregnancy.
* To define the trends of serum uric acid, lipids and xanthine oxidase activity in normotensive and hypertensive pregnancies.
* To determine the ability of the combination of arterial tonometry and endothelial glycocalyx measurement, performed in the two study visits during pregnancy, in predicting the risk of long-term maternal cardiovascular disease.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years
* Single pregnancy
* No previous pregnancies lasting more than 12 weeks
* Participant willing and able to give informed consent for participation in the study

Exclusion Criteria:

* Intermediate-high risk of genetic abnormalities and/or need to perform invasive tests (amniocentesis, villocentesis)
* History of solid organ or hematopoietic stem cell transplantation
* Chronic renal failure (eGFR≤45ml/min/1.73m2)
* Chronic treatment with antihypertensive drugs and/or xanthine oxidase (XO) inhibitors

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2031-09 (Estimated)

PRIMARY OUTCOMES:
Perfused Boundary Region (PBR) | Baseline visit (11/13+6 weeks of pregnancy)
  Micron
Perfused Boundary Region (PBR) | Follow-up visit (24/27+6 weeks of pregnancy)
  Micron
Carotid-femoral pulse wave velocity (cf-PWV) | Baseline visit (11/13+6 weeks of pregnancy)
  m/s
Carotid-femoral pulse wave velocity (cf-PWV) | Follow-up visit (24/27+6 weeks of pregnancy)
  m/s
Number of participants with hypertensive disorders of pregnancy | From date of enrolment until the date of first documented diagnosis of hypertensive disorder of pregnancy, according to the International Society for the Study of Hypertension in Pregnancy Criteria, assessed up to one week after delivery
  Number of participants diagnosed during pregnancy with any hypertensive disorder of pregnancy
Number of participants with preeclampsia | From date of enrolment until the date of first documented diagnosis of preeclampsia, according to the International Society for the Study of Hypertension in Pregnancy Criteria, assessed up to one week after delivery
  Number of participants diagnosed during pregnancy with preeclampsia according to the International Society for the Study of Hypertension in Pregnancy (ISSHP) criteria.

SECONDARY OUTCOMES:
Serum Angiopoietin 1 (ANG-1) | Baseline visit (11/13+6 weeks of pregnancy)
  ng/ml
Serum Angiopoietin 1 (ANG-1) | Follow-up visit (24/27+6 weeks of pregnancy)
  ng/ml
Serum Angiopoietin 2 (ANG-2) | Baseline visit (11/13+6 weeks of pregnancy)
  ng/ml
Serum Angiopoietin 2 (ANG-2) | Follow-up visit (24/27+6 weeks of pregnancy)
  ng/ml
Serum Endothelin-1 (ET-1) | Baseline visit (11/13+6 weeks of pregnancy)
  Serum concentration assessed by ELISA (pg/ml)
Serum Endothelin-1 (ET-1) | Follow-up visit (24/27+6 weeks of pregnancy)
  pg/ml
Serum Intercellular adhesion molecule-1 (ICAM-1) | Baseline visit (11/13+6 weeks of pregnancy)
  ng/ml
Serum Intercellular adhesion molecule-1 (ICAM-1) | Follow-up visit (24/27+6 weeks of pregnancy)
  ng/ml
Serum Vascular Cell Adhesion Molecule-1 (VCAM-1) | Baseline visit (11/13+6 weeks of pregnancy)
  ng/ml
Serum Vascular Cell Adhesion Molecule-1 (VCAM-1) | Follow-up visit (24/27+6 weeks of pregnancy)
  ng/ml
Number of participants with long-term cardiovascular outcomes | Interview 5 years after delivery
  Number of participants diagnosed with stroke, myocardial infarction, heart failure or hospitalized for cardiovascular disease in the 5 years after delivery

OTHER OUTCOMES:
Serum uric acid | Baseline visit (11/13+6 weeks of pregnancy)
  mg/dl
Serum uric acid | Follow-up visit (24/27+6 weeks of pregnancy)
  mg/dl
Serum lipid profile | Baseline visit (11/13+6 weeks of pregnancy)
  HDL-cholesterol (mg/dl), LDL-cholesterol (mg/dl), Triglycerides (mg/dl), Lipoprotein (a) (mg/dl)
Serum lipid profile | Follow-up visit (24/27+6 weeks of pregnancy)
  HDL-cholesterol (mg/dl), LDL-cholesterol (mg/dl), Triglycerides (mg/dl), Lipoprotein (a) (mg/dl)
Xanthine Oxidase Activity | Baseline visit (11/13+6 weeks of pregnancy)
  mU/mL
Xanthine Oxidase Activity | Follow-up visit (24/27+6 weeks of pregnancy)
  mU/mL

CONTACTS AND LOCATIONS:
Overall Officials: Arrigo Francesco Giuseppe Cicero, MD, PhD, Principal Investigator — IRCCS University Hospital of Bologna, Italy. University of Bologna, Italy.
Locations (1):
- Cardiovascular Internal Medicine Unit, IRCCS University Hospital of Bologna, Bologna, Italy, Bologna, Italy

IPD SHARING:
Plan to Share IPD: Yes
All de-identified IPD that underlie results in a publication for all primary and secondary outcome measures will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available after the associated manuscript will be published. No ad-interim analysis is planned before enrollment conclusion.
Access Criteria: Access to IPD can be requested by qualified researchers engaging in independent scientific research, and provided after review and approval of a research proposal and execution of a Data Sharing Agreement (DSA).